CLINICAL TRIAL: NCT01825863
Title: Optimal Postoperative Pain Management by Ultrasound-guided Abdominal Wall Nerve Blockade in Laparoscopic Surgery for Acute Appendicitis - a Randomised Controlled Trial.
Brief Title: Ultrasound-guided Abdominal Wall Nerve Blockade in Laparoscopic Surgery for Acute Appendicitis.
Acronym: BD-TAP APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jens Borglum Neimann, Associate professor, consultant anesthetist, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBH-BDTAP-APP
Record Dates: First submitted 2013-03-27; First posted 2013-04-08 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Appendicitis
Keywords: Laparoscopy; Adult; Nerve block; Ultrasonography
MeSH Terms: conditions — Appendicitis | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active abdominal wall block (Active Comparator): 60ml ropivacaine 0.375% single shot
  Interventions: Drug: Ropivacaine
- Placebo abdominal wall block (Placebo Comparator): 60ml saline 9% single shot
  Interventions: Drug: Saline 9%

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Active abdominal wall block
Drug: Saline 9%
  Arms: Placebo abdominal wall block

SUMMARY:
Acute appendicitis is a common disease and usually occurs within the ages of 10-30 years old." Ten percent of the population will get this disease during a lifetime." At Bispebjerg hospital it is one of the most common acute surgeries performed. Though at Bispebjerg hospital the surgery is only performed on adults as there is no pediatric ward. The surgical technique is primarily laparoscopic surgery, where the patients have their appendix removed while in general anaesthesia. During the last three years Bispebjerg hospital has had an average of 287 patients per year undergoing laparoscopic surgery. From January to the September 2012 a total of 211 patients have had the operation, with 29% having the operation performed during daytime, 48% in the evening and 22% at night. Open appendectomy is only performed in cases where laparoscopic surgery is impossible, this is often due to adhesions, scar tissue from former abdominal surgery or peritonitis. The scars from laparoscopic surgery are usually smaller than that from an open appendectomy, but it gives the patient three smaller scars divided on three abdominal quadrants instead of one larger scar on one quadrant.

The investigators want to conduct a clinical trial with fifty six patients undergoing laparoscopic surgery due to acute appendicitis. The investigators want to find out if it is possible to improve the post-operative pain management within this very large group of patients undergoing acute surgery. In detail, the investigators wish to explore whether the use of the BD-TAP blockade in the abdominal wall on patients undergoing laparoscopic surgery due to acute appendicitis, can anesthetize the patients completely or partially, so they can avoid morphine intake completely or partially during the post-operative phase (12-24 hours). The research project will be a randomized, double-blinded, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patients undergoing diagnostic laparoscopy for acute appendicitis
* American Society of Anaesthesiology group 1-3
* General Anaesthesia

Exclusion Criteria:

* Inability to cooperate
* Inability to understand and talk danish
* Allergic to ropivacaine
* Drug and alcohol abuse
* Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC), 0-12 hours, numerical rating score-pain-(NRS)0-10 | 0-12 hours postoperatively
  Pain score (NRS) assessed when sitting up 0-12 hours postoperatively. AUC is calculated over a time frame of 0-12 hours.

SECONDARY OUTCOMES:
Area under the curve (AUC), 0-12 hours postoperatively, numerical rating score - pain-(NRS) 0-10 | 0-12 hours postoperatively
  NRS 0-10 is assessed 0-12 hours postoperatively. AUC is calculated 0-12 hours postoperatively.
Morphine consumption postoperatively | 0-12 hours postoperatively
  Morphine consumption postoperatively registered from the patient controlled analgesia (PCA) pump.
Length of stay (LOS) in the postanesthesia care unit (PACU) | Time from arrival in PACU to time of departure (measured in minutes)
Side effects related to morphine consumption | 0-12 hours postoperatively
  Side effects recorded: nausea and vomiting
Time to first mobilisation 0-12 hours postoperatively | 0-12 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Tanggaard, research year fellow, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of anaesthesiology, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Borglum J, Jensen K, Christensen AF, Hoegberg LC, Johansen SS, Lonnqvist PA, Jansen T. Distribution patterns, dermatomal anesthesia, and ropivacaine serum concentrations after bilateral dual transversus abdominis plane block. Reg Anesth Pain Med. 2012 May-Jun;37(3):294-301. doi: 10.1097/AAP.0b013e31824c20a9. PMID 22476239